CLINICAL TRIAL: NCT06076772
Title: Palbociclib Induced Neutropenia; Risk Factors and Treatment Outcome in Metastatic Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa I Mekkawy, Principal Investigator, Assiut University
Other Study IDs: Palbociclib
Record Dates: First submitted 2023-09-18; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: cases developed neutropenia Grade 0-2 with palbociclib administration
  Interventions: Drug: Palbociclib
- 2: cases developed neutropenia Grade 3-4 with palbociclib administration
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — The investigator will follow the patients after starting treatment to follow and observe the outcome of the treatment side effects and risk factors
  Other Names: Other drugs (hormonal treatment)+ denosumab

SUMMARY:
Aim of the study to assess the neutropenia induced by Palbociclib in patient receiving Palbociclib in combination with hormonal treatment as first-line therapy in metastatic hormone receptor- positive HER2 negative breast cancer. To evaluate the risk factors for occurrence of neutropenia and treatment outcome as 2 years PFS and OS.

DETAILED DESCRIPTION:
Palbociclib is an orally active cyclin-dependent kinase (CDK) and is considered the standard treatment for hormone receptor (HR)-positive, (HER) negative metastatic breast cancer.

The PALOMA studies' showed improvement in progression-free survival (PFS) compared to endocrine therapy alone but a non-significant trend towards improved overall survival (OS).

MONALEESA and MONARCH suggest significantly improved OS with the addition of CDK inhibition.

Neutropenia is considered the dose-limiting and most frequent adverse effect of CDK inhibitors resulting in frequent dose reductions and treatment interruptions that are potentially associated with a lack of efficiency. Grade III/IV neutropenia rates were 62-66% in the PALOMA studies.

Some studies investigated the risk factors for the development of palbociclib-induced neutropenia. One concluded that no concomitant use of statins and high BMI were identified as significant predictors for the development of palbociclib-induced neutropenia. and another study also concluded that low baseline ANC, WBC, PLT, and BSA were associated with early grade III/IV neutropenia.

Regarding treatment outcome, two Phase Two clinical trials concluded that the treatment-related neutropenia in the first two cycles was significantly and independently associated with prolonged PFS, suggesting that neutropenia may be a useful pharmacodynamic marker to guide individualised palbociclib dosing.

However, another study concluded that limited dose modification may lead to longer PFS, without increasing toxicity, than the conventional dose scheme.

A study of variable risk factors and treatment outcomes for palbociclib-induced neutropenia will be useful for careful monitoring leading to adapted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological pathological confirmation of primary breast cancer or metastatic disease.
* Hormonal receptor-positive, HER2 negative.
* Metastatic breast cancer at presentation (Den novo) or recurrent.
* Patients did not receive any previous systemic therapy for metastatic disease.
* Performance status (ECOG) 0-2.

Exclusion Criteria:

* Patient with co-morbidity
* Pregnant and breast lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient receiving Palbociclib in combination with hormonal treatment as first-line therapy in metastatic hormone receptor- positive HER2 negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Investigator will evaluate the patients and treatment characters in counts and percentage of developing high-grade neutropenia induced by palbociclib. | 2 years
  Investigator will record the patients and treatment characters in counts and percentage that associated with the occurrence of high-grade neutropenia. And then will compare the characters differences in patients with and without high grade neutropenia by uninitiated and multivariate statistical analysis.
assess treatment outcome as a progression free survival for palbociclib in patient with neutropenia | 2 years
  Measure the progression free survival
assess treatment outcome as overall survival for palbociclib in patient with neutropenia | 2 years
  Measure the overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Imam Ahmed, Al Madīnah, AL, Saudi Arabia

REFERENCES:
- [Background] Kim SG, Kim MH, Park S, Kim GM, Kim JH, Kim JY, Park HS, Park S, Park BW, Kim SI, Ji JH, Jeong J, Shin K, Lee J, Kim HD, Jung KH, Sohn J. Efficacy of Limited Dose Modifications for Palbociclib-Related Grade 3 Neutropenia in Hormone Receptor-Positive Metastatic Breast Cancer. Cancer Res Treat. 2023 Oct;55(4):1198-1209. doi: 10.4143/crt.2022.1543. Epub 2023 Apr 11. PMID 37054718
- [Background] McAndrew NP, Dickson MA, Clark AS, Troxel AB, O'Hara MH, Colameco C, Gallager M, Gramlich K, Zafman K, Vaughn D, Schwartz GK, O'Dwyer PJ, DeMichele A. Early treatment-related neutropenia predicts response to palbociclib. Br J Cancer. 2020 Sep;123(6):912-918. doi: 10.1038/s41416-020-0967-7. Epub 2020 Jul 9. PMID 32641862
- [Background] Lavery L, DiSogra K, Lea J, Trufan SJ, Symanowski JT, Roberts A, Moore DC, Heeke A, Pal S. Risk factors associated with palbociclib-induced neutropenia in patients with metastatic breast cancer. Support Care Cancer. 2022 Dec;30(12):9803-9809. doi: 10.1007/s00520-022-07400-z. Epub 2022 Oct 19. PMID 36260177
- [Background] Kanbayashi Y, Sakaguchi K, Ishikawa T, Takayama K, Taguchi T. Predictors for development of palbociclib-induced neutropenia in breast cancer patients as determined by ordered logistic regression analysis. Sci Rep. 2021 Oct 8;11(1):20055. doi: 10.1038/s41598-021-99504-5. PMID 34625634
- [Background] Lee Y, Lee D, Seo I, Chae H, Sim SH, Lee KS, Gwak HS. Risk Factors for Palbociclib-Induced Early Developing Neutropenia in Patients with Hormone Receptor-Positive Metastatic Breast Cancer. Cancers (Basel). 2023 May 18;15(10):2810. doi: 10.3390/cancers15102810. PMID 37345147
- [Background] Vazquez L, Arnaud A, Grenier J, Debourdeau P. [Patients treated with palbociclib and endocrine therapy for metastatic breast cancer: Can we predict the occurrence of severe early hematological toxicity?]. Bull Cancer. 2021 May;108(5):544-552. doi: 10.1016/j.bulcan.2021.01.007. Epub 2021 Apr 2. French. PMID 33820647